CLINICAL TRIAL: NCT06006559
Title: A Randomized, Participant- and Investigator-blinded, Placebo-controlled, Parallel Group Study to Assess the Efficacy, Safety and Pharmacokinetics of EYU688 in Patients With Dengue Fever
Brief Title: A Study to Assess the Efficacy, Safety and Pharmacokinetics of EYU688 in Patients With Dengue Fever
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEYU688A12201
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Dengue
Keywords: Dengue; EYU688
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EYU688 (Experimental): EYU688 administered by oral route
  Interventions: Drug: EYU688
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EYU688 — EYU688 administered by oral route
  Arms: EYU688
Drug: Placebo — Matching placebo administered orally as capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the effect on dengue viral load, fever clearance time as well as on clinical signs and symptoms with the treatment of EYU688 compared with placebo in patients with dengue fever.

DETAILED DESCRIPTION:
This is a randomized, participant- and investigator- blinded, placebo-controlled study to investigate the efficacy and safety of EYU688 administered orally in patients with dengue fever.

Due to the different PK sampling schedules applied, the study consists of two cohorts run in parallel (intensive PK [cohort 1] and sparse PK sampling [cohort 2]).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 60 years old (inclusive).
* History or presence of fever (≥ 38°C). At least one of the following criteria indicating dengue infection:
* Nausea or vomiting.
* Presence of rash, aches or pains including headache, muscle or joint pain.
* Onset of fever ≤ 48 hours prior to treatment start.
* Positive test on dengue fever.

Exclusion Criteria:

* Participants with any of abnormalities of clinical laboratory parameters.
* Usage of any anticoagulant drugs.
* Current significant medical conditions or illness that the investigator considers should exclude the participants, especially those that require continuation of other medications likely to have an interaction with the study drug.
* Pregnant or nursing (lactating) women.
* Clinical signs and symptoms for severe dengue according to Dengue Guideline (WHO 2009) at screening.
* Participants with any of the following abnormalities of clinical laboratory parameters at screening:

  * Hemoglobin <12.0 g/dL in males; <11.0 g/dL in females
  * Hematocrit >52 % in males; >46 % in females
  * Absolute neutrophil count <1500/μL
  * Platelet count <80,000/mm3
  * Creatinine >165 μmol/L in males; >130 μmol/L in females
  * Serum creatine kinase > 600 U/L
  * ALT, AST levels more than 1.5X upper limit of normal (ULN)
  * Total bilirubin >24 μmol/L
* Usage of PPIs (proton pump inhibitor) which could affect absorption of EYU688 due to stomach pH value increase up to 48 hours prior to screening.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 4 days after stopping of investigational drug.
* History or long-QT syndrome, or clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening:

  * QTcF > 450 msec (males)
  * QTcF > 460 msec (females)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Viremia reduction (viral load reduction (VLR) on log scale) at 48 hours post treatment start | From predose to 48 hours post treatment start
  Efficacy assessment of EYU688. It will allow to quantify the viremia reduction at 48 hours post treatment start from baseline.

SECONDARY OUTCOMES:
Time from fever onset to start of the first 48 hours period during which the oral temperature remained below 37.5℃ | From fever onset to Day 15
  Efficacy assessment of EYU688. It will allow to assess the time needed between fever onset and defervescence.
Time from fever onset to the first of two consecutive negative viremia by PCR | From fever onset to Day 15
  Efficacy assessment will allow to assess the viremia kinetic from treatment start to Day15
Area under the log-transformed viremia curve (AUC) from the first dose to Day 15 | From fever onset to Day 15
  Efficacy assessment will allow to assess the viremia kinetic from treatment start to Day 15
Changes of viral load over time | From baseline to Day 15
  Efficacy assessment will allow to assess the viremia kinetic from treatment start to Day15
Incidence and severity of Adverse Events (AEs) | From inclusion to Day 15
  Incidence and severity of AEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Incidence and severity of Serious Adverse Events (SAEs) | From inclusion to Day 35
  Incidence and severity of SAEs by treatment group
Change of white blood cell count over time from baseline | From baseline to Day 15
  Assessment of safety and tolerability of EYU688
Change of platelet count over time | From baseline to Day 15
  Assessment of safety and tolerability of EYU688
Change of hematocrit level and percentage increase from baseline over time | From baseline to Day 15
  Assessment of safety and tolerability of EYU688
Change of AST, ALT levels over time | From baseline to Day 15
  Assessment of safety and tolerability of EYU688
No warning signs by day 7 of fever onset | From inclusion to Day 15
  Assessment of the dengue fever clinical evolution under EYU688
Diagnosis of severe dengue fever | From inclusion to Day 15
  Assessment of the dengue fever clinical evolution under EYU688
Diagnosis of dengue hemorrhagic fever (DHF) | From inclusion to Day 15
  Assessment of the dengue fever clinical evolution under EYU688
Plasma leakage | From inclusion to Day 15
  Assessment of the dengue fever clinical evolution under EYU688
Requiring fluid infusion | From inclusion to Day 15
  Assessment of the dengue fever clinical evolution under EYU688
Time from fever onset to clinical recovery | From fever onset to Day 15
  Assessment of the dengue fever clinical evolution under EYU688
PK parameter (Cmax) | From Day 1 to Day 6
  Pharmacokinetic assessment of EYU688 in dengue fever patients
PK parameter (Tmax) | From Day 1 to Day 6
  Pharmacokinetic assessment of EYU688 in dengue fever patients
PK parameter (partial AUCs) | From Day 1 to Day 6
  Pharmacokinetic assessment of EYU688 in dengue fever patients
PK concentrations following multiple doses | From Day 1 to Day 6
  Pharmacokinetic assessment of EYU688 in dengue fever patients

CONTACTS AND LOCATIONS:
Locations (22):
- Brazil (5):
  - Novartis Investigative Site, Manaus, Amazonas
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Sorocaba, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
- India (5):
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
- Malaysia (5):
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Seberang Jaya, Pulau Pinang
  - Novartis Investigative Site, Miri, Sarawak
  - Novartis Investigative Site, Kuala Selangor
- Novartis Investigative Site, Singapore, Singapore
- Vietnam (3):
  - Novartis Investigative Site, Haiphong
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.